CLINICAL TRIAL: NCT05780216
Title: Mindfulness and Psychedelics: A Combined Neurophenomenological and Pharmacological Approach to the Characterization of Mindfulness States in Experienced Meditators
Brief Title: Mindfulness and Psychedelics
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Milan Scheidegger (Other)
Collaborators: University Medical Center Freiburg (Other)
Responsible Party: Sponsor-Investigator, Milan Scheidegger, Principal Investigator, Junior Group Leader, Senior Physician, Psychiatric University Hospital, Zurich
Organization: Psychiatric University Hospital, Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: DMT-HAR-MED
Record Dates: First submitted 2023-02-23; First posted 2023-03-22 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Healthy Participants
Keywords: DMT; harmine; pharmahuasca; ayahuasca; healthy participants; meditation; group retreat; mindfulness
MeSH Terms: interventions — N,N-Dimethyltryptamine; Harmine

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, placebo-controlled, between-subjects study design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DMT and harmine (Experimental): This arm comprises the following interventions:
  * Mindfulness Intervention in the course of the meditation group retreat
  * Administration of DMT + harmine (moderate-high dose)
  Interventions: Drug: DMT + harmine
- Placebo (Placebo Comparator): This arm comprises the following interventions:
  * Mindfulness Intervention in the course of the meditation group retreat
  * Administration of Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DMT + harmine — The intervention used in this study is a combination of the two main ingredients of ayahuasca, DMT (N,N-dimethyltryptamine) and harmine in purified form.
  Arms: DMT and harmine
Drug: Placebo — The placebo consists of pharmaceutically inactive ingredients and additional flavors, and is organoleptically hardly distinguishable from the verum.
  Arms: Placebo

SUMMARY:
The investigators are doing this project to investigate potential neurophysiological synergy effects between mindfulness meditation and psychedelics. Previous studies have found that both mindfulness and psychedelics like psilocybin modulate neural activity and connectivity of the same brain network. However, little is known about the potential interactions between mindfulness meditation and psychedelics. The indigenous plant preparation "Ayahuasca" is particularly interesting for the combination with mindfulness meditation. It contains two components, N,N-dimethyltryptamine (DMT) and harmine, which are very similar to the body's own messenger substance serotonin and increase its effect in the body. The investigators would now like to find out how these corresponding networks change in experienced meditators after DMT/Harmine-enhanced mindfulness meditation and how this affects their subjective experience. For this functional MRI imaging will be performed, as well as psychometric assessments and detailed experiential interviews before and after a three-day meditation retreat. Participants will be randomly assigned to one of two groups. One group receives DMT and harmine during the sitting meditation on the second day, the other group receives a corresponding placebo. Neither the participants nor the investigator know who will receive a placebo or the combination of DMT/harmine on the day of the experiment. The pre- and post-measurements of the MRI imaging and psychometric questionnaires of the DMT/Harmine group are compared with those of the placebo control group. By examining the synergistic effects of mindfulness meditation and DMT/harmine, the aim of this study is to contribute to a comprehensive understanding of the neurophenomenology of rare and inaccessible phenomena of consciousness.

ELIGIBILITY:
Inclusion Criteria:

* Willing and capable to give informed consent for the participation in the study after it has been thoroughly explained
* Not more than little experience with psychedelic substances
* Experience in Buddhist meditation: participants have a minimum of 1000 hours of lifetime formal meditation practice, e.g. Mahayana (Zen) Theravada (Vipassana) Buddhism or Mahamudra/Dzogchen as primary meditation background, familiarity with longer periods of meditation in a retreat setting.
* Body mass index (BMI) between 18.5 and 35
* Willing to refrain from drinking alcohol during the retreat and caffeinated drinks at the testing days and from consuming psychoactive substances or other medications for 2 weeks before testing days and for the duration of the study
* Able and willing to comply with all study requirements
* Informed consent form was signed
* Good knowledge of the German language
* Participant informs study physicians / project scientists about simultaneous treatment or therapy with other physicians and about current intake of psychotropic substances or medication
* Women of childbearing potential are required to use effective, established contraception, such as oral, injected or implanted hormonal methods of contraception, placement of an intrauterine device (IUD) or intrauterine system (IUS), barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository

Exclusion Criteria:

* Previous significant adverse response to a hallucinogenic drug or to a mindfulness intervention (e.g. meditation retreat)
* Participation in another study where pharmaceutical compounds will be given
* Presence of Axis I affective, anxiety, or dissociative disorders
* Present or antecedent diagnosis of bipolar disorder (I, II, not otherwise specified), schizophrenia, schizoaffective disorder, psychosis, or other disorders from the psychotic spectrum
* First-degree relatives with present or antecedent schizophrenia, schizoaffective disorder, or bipolar disorder type I
* History of head trauma, seizures, cancer, or cerebrovascular accidents
* Recent cardiac or brain surgery
* Current abuse of medication or psychotropic substances (including nicotine addiction) according to SCID I criteria
* Presence of major internal or neurological disorders (including sepsis, pheochromocytoma, thyrotoxicosis, drug-induced fibrosis, familiar or basilar artery migraine)
* Cardiovascular disease (hypertonia, coronary artery disease, heart insufficiency, myocardial infarction, coronary spastic angina)
* Peripheral vascular disease (thromboangiitis obliterans, luetic arteritis, severe arteriosclerosis, thrombophlebitis, Raynaud's disease)
* Cerebrovascular disease (e.g. stroke, intracranial bleeding / hemorrhage, intracranial aneurysm)
* Serious abnormalities in ECG or blood count/chemistry
* Liver or renal or pulmonary disease
* Pregnant or breastfeeding women (a urine pregnancy test will be done for all women capable of bearing children)
* Inability to lie still for about 60 minutes (e.g. because of sneezing, itching, tremor, pain)
* Left-handedness
* MRI-exclusion criteria: Metal parts in the body (piercings, brain aneurysm clip, implanted neural stimulator/cardiac pacemaker/defibrillator/Swan Ganz catheter/insulin pump, cochlear implant); metal shrapnel or bullet, ocular foreign body (e.g. metal shavings); current or previous job in metalworking industry
* Claustrophobia
* Current use of medications with significant interaction potential with MAOI (e.g. antidepressants, antipsychotics, psychostimulants, dopaminergic/serotonergic agents, anticonvulsants);
* high risk of adverse emotional or behavioral reaction based on investigator's clinical evaluation (e.g. evidence of serious personality disorder, serious current stressors, lack of social support).

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2023-08-05 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Functional brain connectivity changes in response to DMT-enhanced mindfulness in experienced meditators (rs-fMRI) | fMRI recordings 1 day before the group meditation retreat - fMRI recordings 1 day after the group meditation retreat
  The primary endpoint of this present study is to test functional brain connectivity at rest and during meditation in response to DMT-enhanced mindfulness in experienced meditators. More specifically, the present study aims at assessing the impact of DMT-enhanced mindfulness on the attenuation of Default Mode Network (DMN) activity and connectivity with fMRI recordings before and after a group meditation retreat using SVA and ICA analyses.

SECONDARY OUTCOMES:
Psychometric changes in response to DMT-enhanced mindfulness in experienced meditators | Baseline - Retreat Day 2 (i.e. study day with pharmacological intervention) - Retreat Day 3
  Measures of drug-induced altered states of consciousness:
  Mystical Experience Questionnaire (minimum value = 0; maximum value = 5; higher scores indicate individual mystical experiences)
Psychometric changes in response to DMT-enhanced mindfulness in experienced meditators | Retreat Day 1 - Retreat Day 2 (i.e. study day with pharmacological intervention) - Retreat Day 3
  Measures of drug-induced altered states of consciousness:
  Visual Self-Transcendence Scale (minimum value = 1; maximum value = 7; higher scores indicate higher self-transcendence)
Psychometric changes in response to DMT-enhanced mindfulness in experienced meditators | Baseline - Retreat Day 2 (i.e. study day with pharmacological intervention) - Retreat Day 3
  Measures of drug-induced altered states of consciousness:
  Non-dual Awareness Dimensional Assessment Scale-State (visual analog scale; minimum value = 0; maximum value = 10)
Psychometric changes in response to DMT-enhanced mindfulness in experienced meditators | Follow-up 1 month after the group meditation retreat
  Measures of drug-induced altered states of consciousness:
  Persisting Effects Questionnaire (minimum value = no change [1]; maximum value = very strong change [5]; higher scores indicate greater change)
Psychometric changes in response to DMT-enhanced mindfulness in experienced meditators | Baseline - Study Day with pharmacological intervention - 1 day after the group retreat - Follow-up 1 week after the group meditation retreat
  Mindfulness & Compassion:
  Toronto Mindfulness Scale (minimum value = 0; maximum value = 4; higher scores indicate greater mindfulness) Meditation Depth Questionnaire (minimum value = 0; maximum value = 4) Sussex-Oxford Compassion Scale (minimum value = 0; maximum value = 4)
Psychometric changes in response to DMT-enhanced mindfulness in experienced meditators | Baseline - Study Day with pharmacological intervention - 1 day after the group retreat - Follow-up 1 week after the group meditation retreat
  Connectedness:
  Watts Connectedness Scale (visual analog scale; minimum value = 0; maximum value = 100)
Psychometric changes in response to DMT-enhanced mindfulness in experienced meditators | Baseline - 1 day after the group retreat - Follow-up 1 week after the group meditation retreat
  Mindfulness:
  Freiburg Mindfulness Inventory (minimum value = 1; maximum value = 4; higher scores indicate greater mindfulness)
Psychometric changes in response to DMT-enhanced mindfulness in experienced meditators | Baseline - Study Day with pharmacological intervention - Retreat Day 3 - 1 day after the group meditation retreat - Follow-up 1 week after the group meditation retreat
  Gratitude:
  Gratitude Questionnaire (minimum value = 1; maximum value = 7)
Psychometric changes in response to DMT-enhanced mindfulness in experienced meditators | Retreat Day 1 - Retreat Day 2 (i.e. study day with pharmacological intervention) - Retreat Day 3
  Psychological Insights:
  Psychological Insight Scale (visual analog scale: left = not more than before; right = very much more than before)
Psychometric changes in response to DMT-enhanced mindfulness in experienced meditators | 1 day before the group meditation retreat -1 day after the group meditation retreat - Follow-up 1 week after the group meditation retreat
  Psychological Flexibility:
  Psy-Flex Questionnaire (minimum value = 1; maximum value = 5; higher scores indicate greater psychological flexibility)
Phenomenological reports in response to DMT-enhanced mindfulness in experienced meditators | Within 24 hours after drug administration - Follow-up 1 month after the group meditation retreat
  Microphenomenological and semi-structured qualitative interviews
Incidence of Treatment-Emergent Adverse Events | On study days with pharmacological intervention (at baseline, 30, 60, 90, 120, 180, 240, and 360 min after drug administration)
  Frequency of occurence of treatment-related adverse events as assessed by CTCAE v5.0
EmpaToM (fMRI task) | fMRI recordings 1 day before the group meditation retreat - fMRI recordings 1 day after the group meditation retreat
  The EmpaToM is a validated fMRI test paradigm to assess emotional valence, compassion or empathy and theory of mind
Mediating Variables | Baseline - Study Day with pharmacological intervention - 1 day after group meditation retreat - Follow-up 1 week after the group meditation retreat
  Personality Type:
  Ten-Item Personality Inventory (minimal value =1; maximal value = 7)
Mediating Variables | Baseline
  Personality Type:
  Affective Neuroscience Personality Scale (minimum value = 1; maximum value = 4)
Mediating Variables | Baseline - Study Day with pharmacological intervention - Retreat Day 3 - Follow-up 1 week and 1 month after the group meditation retreat
  Meditation Motivation (single-choice) & Intention (visual analog scale)
Mediating Variables | Immediately before the pharmacological intervention
  Expectations (minimal value = 0; maximal value = 4)

CONTACTS AND LOCATIONS:
Overall Officials: Milan Scheidegger, MD, PhD, Principal Investigator — Psychiatric University Hospital, Zurich
Locations (1):
- Psychiatric University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
Only anonymized, quantitative neurophysiological and behavioral data can be shared upon publication according to the FAIR data principles. Qualitative interview data are sensitive and cannot be shared due to confidentiality reasons.

REFERENCES:
- [Derived] Meling D, Egger K, Aicher HD, Jareno Redondo J, Mueller J, Dornbierer J, Temperli E, Vasella EA, Caflisch L, Pfeiffer DJ, Schlomberg JT, Smallridge JW, Dornbierer DA, Scheidegger M. Meditating on psychedelics. A randomized placebo-controlled study of DMT and harmine in a mindfulness retreat. J Psychopharmacol. 2024 Oct;38(10):897-910. doi: 10.1177/02698811241282637. Epub 2024 Sep 27. PMID 39340164